CLINICAL TRIAL: NCT03102502
Title: Study of the Effects of Enhanced External Counterpulsation on Vascular Hemodynamics and Status
Brief Title: Impact of Enhanced External Counterpulsation on Vascular Hemodynamics and Status
Acronym: EECPVHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yan Zhang, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EECP- 2
Record Dates: First submitted 2017-03-31; First posted 2017-04-05 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Atherosclerosis; Vascular Endothelium; Counterpulsation, External
MeSH Terms: conditions — Coronary Disease; Atherosclerosis | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Parallel: Patiants with coronary heart disease are assigned to two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced External Counterpulsation (Experimental): Patients receive a total of 35-36 hours of EECP treatment on top of guideline- driven standard medical therapy for coronary heart disease, 1-hour sessions every day over a 7-week period.
  Interventions: Device: EECP; Drug: Medical therapy
- Control (Active Comparator): Patients receive guideline- driven standard medical therapy for 7 weeks without Enhanced External Counterpulsation intervention.
  Interventions: Drug: Medical therapy

INTERVENTIONS:
Device: EECP — Enhanced external counterpulsation (EECP) is a technique for assisting the circulation by decreasing the afterload of the left ventricle and augmenting the diastolic pressure externally by applying a negative pressure to the lower extremities during cardiac systole. EECP therapy is done by sequential inflation of 3 sets of cuffs wrapped around the lower extremities during diastole and deflation of the cuffs during systole. EECP enhances the aortic diastolic blood flow and coronary perfusion, leading to increased arterial wall shear stress in a pulsatile manner.
  Other Names: Enhanced External Counterpulsation
  Arms: Enhanced External Counterpulsation
Drug: Medical therapy — Guideline- driven standard medical treatment including statins,antiplatelet drugs（aspirin or Clopidogrel ）, anti-ischemic drugs （Nitroglycerin）
  Other Names: Guideline- driven medical therapy

SUMMARY:
The present study aimed to investigated the effect of Enhanced External Counterpulsation (EECP) on vascular hemodynamics and atherosclerosis, and the underlying shear stress related mechanisms

DETAILED DESCRIPTION:
Patients with coronary heart disease will be randomized into two groups: standard medical treatment and standard medical treatment plus EECP intervention. Hemodynamic parameters, vascular status and function will be measured.

ELIGIBILITY:
Inclusion Criteria:

* More than 50% stenosis of left main trunk and 3 epicardial coronary arteries and their large branches showed by coronary angiography
* Or history of myocardial infarction
* Or history of prior revascularization
* Signed informed consent to participate in the study

Exclusion Criteria:

* Clinically significant valvular heart disease
* Aortic aneurysm
* Congenital heart disease
* Acute myocarditis
* Arrythmias significantly interfere with the triggering of the EECP device
* History of cerebral hemorrhage
* Hemorrhagic disease
* Lower limb infection, phlebitis
* Deep venous thrombosis
* Malignant disease
* INR > 2.5
* Uncontrolled hypertension, defined as SBP > 180mmHg or DBP > 110mmHg
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Change in blood flow velocity | At baseline, during EECP and week 7 (post intervention)
  Change from baseline in blood flow velocity measured by color Doppler ultrasound system

SECONDARY OUTCOMES:
Change in vascular endothelial function | At baseline and week 7 (post intervention)
  Change from baseline in flow- mediated dilation (FMD) accessed by color Doppler ultrasound system
Change in atherosclerosis | At baseline and week 7 (post intervention)
  Change from baseline in atherosclerosis : plaque of common carotid artery, carotid intima- media thickness, pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M. D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Zhensheng Zheng, M. D., Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat- sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchanda A, Soran O. Enhanced external counterpulsation and future directions: step beyond medical management for patients with angina and heart failure. J Am Coll Cardiol. 2007 Oct 16;50(16):1523-31. doi: 10.1016/j.jacc.2007.07.024. Epub 2007 Oct 1. PMID 17936150
- [Background] Nichols WW, Estrada JC, Braith RW, Owens K, Conti CR. Enhanced external counterpulsation treatment improves arterial wall properties and wave reflection characteristics in patients with refractory angina. J Am Coll Cardiol. 2006 Sep 19;48(6):1208-14. doi: 10.1016/j.jacc.2006.04.094. Epub 2006 Aug 28. PMID 16979007
- [Background] Braith RW, Conti CR, Nichols WW, Choi CY, Khuddus MA, Beck DT, Casey DP. Enhanced external counterpulsation improves peripheral artery flow-mediated dilation in patients with chronic angina: a randomized sham-controlled study. Circulation. 2010 Oct 19;122(16):1612-20. doi: 10.1161/CIRCULATIONAHA.109.923482. Epub 2010 Oct 4. PMID 20921442
- [Background] Zhang Y, He X, Chen X, Ma H, Liu D, Luo J, Du Z, Jin Y, Xiong Y, He J, Fang D, Wang K, Lawson WE, Hui JC, Zheng Z, Wu G. Enhanced external counterpulsation inhibits intimal hyperplasia by modifying shear stress responsive gene expression in hypercholesterolemic pigs. Circulation. 2007 Jul 31;116(5):526-34. doi: 10.1161/CIRCULATIONAHA.106.647248. Epub 2007 Jul 9. PMID 17620513